CLINICAL TRIAL: NCT00800969
Title: Prospective Evaluation of the Preoperative Lymph Node Staging in Patients With Cancer of the Esophagogastric Junction and Stomach
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: VIS-UGI-1
Record Dates: First submitted 2008-11-28; First posted 2008-12-03 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Adenocarcinoma; Stomach Cancer; Cancer of Esophagogastric Junction
Keywords: Adenocarcinoma of the stomach and esophagogastric junction
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- all patients (Other): all patients with Adenocarcinoma
  Interventions: Procedure: FDG-PET-CT

INTERVENTIONS:
Procedure: FDG-PET-CT — Radiologic standard procedure

SUMMARY:
This prospective study includes patients with histologically proven cancer of the esophagogastric junction (Siewert Type II and III) and the stomach. Aim of the study is to evaluate the accuracy of PET-CT for the preoperative assessment of lymph node metastasis. The evaluation includes a combination with standard diagnostic tools (endoluminal ultrasound, CT and diagnostic laparoscopy prior to neoadjuvant therapy). Standardized D2-lymphadenectomy is performed and individual lymph node stations (Nr 1-12 according to the Japanese classification) are histopathologically examined. Furthermore we evaluate the role of the PET-CT for early metabolic response evaluation in patients receiving neoadjuvant chemotherapy.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* Histological prove of adenocarcinoma of the stomach.

Exclusion criteria:

* Recurrent gastric carcinoma
* No informed consent
* Previous malignancy (exception: thyroid, bladder in situ, Cervix in situ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of PET-CT | preoperative

CONTACTS AND LOCATIONS:
Overall Officials: Kuno Lehmann, MD, Principal Investigator — University Hospital Zurich, Visceral surgery
Locations (1):
- Zurich, Switzerland